CLINICAL TRIAL: NCT04316013
Title: Volatile Anaesthesia and Perioperative Outcomes Related to Cancer: the VAPOR-C Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not meeting recruitment timelines
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Australian and New Zealand College of Anaesthetists (Other); Victorian Comprehensive Cancer Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18/044
Record Dates: First submitted 2020-01-22; First posted 2020-03-20 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Colonic Cancer; Rectal Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Intervention Model Description: This is an event-driven, international multicentre, randomised controlled trial with a 2x2 factorial design. Patients with stage I-III colorectal cancer or stage I-IIIa NSCLC are eligible and will be randomised in the ratio of 1:1:1:1 using permuted block randomisation with stratification by cancer type (Colon, Rectal or NSCLC), and by site to receive either 1) sevoflurane maintenance anaesthesia and lidocaine infusion or 2) sevoflurane maintenance anaesthesia; or 3), propofol maintenance anaesthesia and lidocaine infusion or 4), propofol maintenance anaesthesia .
Who Masked: Participant
Masking Description: The propofol-TIVA/sevoflurane element of each arm will have a single blind (patient blinded), as the administering anesthesiologist cannot be blinded to allocation. The lidocaine infusion or no lidocaine infusion element of each ARM will be blinded to the patient . The anaesthetic team and research team caring for the patient will not be blinded to the lidocaine infusion/no lidocaine infusion element of the randomisation ARM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- A (Active Comparator): Sevoflurane + intravenous lidocaine
  Interventions: Drug: Sevoflurane; Drug: Lidocaine IV
- B (Active Comparator): Sevoflurane
  Interventions: Drug: Sevoflurane
- C (Active Comparator): Propofol TIVA + intravenous lidocaine
  Interventions: Drug: Propofol; Drug: Lidocaine IV
- D (Active Comparator): Propofol TIVA
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Inhaled anaesthetic used for maintenance of anaesthesia, dosed as per standard practice
  Arms: A; B
Drug: Propofol — Intravenous anaesthetic used for induction and maintenance of anaesthesia
  Arms: C; D
Drug: Lidocaine IV — 1.5mg/kg loading dose over 20 minutes, followed by an infusion of 2mg/kg/hr up to 4 hours and 1.5mg/kg/hour thereafter. Bolus and maintenance dosages of lidocaine will be per actual body weight and capped at a maximum of 100 kg.
  Arms: A; C

SUMMARY:
VAPOR-C is a randomised study of the impact of IV versus inhaled anaesthesia (propofol versus sevoflurane) and lidocaine versus no lidocaine on duration of disease free survival inpatients with either colorectal or non small cell lung cancer.

DETAILED DESCRIPTION:
VAPOR-C is a pragmatic, event-driven, randomised controlled trial, with a single blind 2x2 factorial design for sevoflurane/propofol and for intravenous lidocaine infusion / no lidocaine infusion.

This trial is designed to test for superiority in disease free survival (DFS) of propofol (total intravenous anaesthesia -TIVA) over sevoflurane (inhalational volatile anaesthesia) and intravenous lidocaine over no lidocaine in patients undergoing surgery for colorectal or non small cell lung cancer (NSCLC). The combination of two cancer types will help address the need to demonstrate the effects of anaesthetic technique across cancers to inform generalisable anaesthesia guidelines. Both NSCLC and colorectal cancer are important for this study due to high incidence rate, many longer-term survivors, and importantly the high risk of local or distant recurrence despite complete surgical resection. In addition, the study will collect additional data in a nested cohort related to the exploratory objectives.

The study aims to recruit 3,500 patients in Australia, New Zealand, Canada, United States and Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older at screening
2. Has provided written informed consent for the trial
3. Patient with American Joint committee on Cancer (AJCC) 8th edition Stage I-III colorectal cancer or Stage I-IIIa NSCLC, as confirmed by histological or cytological diagnosis. In cases where a histological diagnosis is not possible, suspected diagnosis through imaging techniques is acceptable.
4. Patient has an American Society of Anaesthesiologists (ASA) score of 1 to 3
5. Scheduled to receive elective, surgical resection with curative intent
6. Surgery expected to last ≥2 hours and expected to require ≥2 nights hospital stay
7. Able to comply with protocol requirements and follow-up procedures

Exclusion Criteria:

1. Confirmed or suspected allergy to propofol, sevoflurane or intravenous lidocaine
2. Patient with significant liver disease (with elevated International Normalised Ratio (INR) or bilirubin and/or low albumin; i.e. Childs-Pugh Score >Class A;
3. Patient at personal or familial risk of malignant hyperthermia or porphyria
4. Patient with a history of other malignancies within the past 5 years. However, patients with malignancies managed with curative therapy and considered to be at low risk of recurrence such as treated skin basal cell carcinoma, squamous cell carcinoma, malignant melanoma ≤1.0mm without ulceration, localised thyroid cancer, cervical carcinoma in situ or prior malignancies with high likelihood of cure (e.g. low grade prostate and breast cancer) may be included in the study
5. Patient has distant metastases
6. Patient with an actual body weight less than 45kg
7. Patients taking the following drugs that are moderate-strong inhibitors of the CYP1A2 and CYP3A4 metabolic pathways within 72 hours prior to surgery: Antibiotics - 'mycin' class: Clarithromycin, Telithromycin, Azithromycin, Erythromycin Antibiotics - 'floxacin' class Ciprofloxacin (exception: can be used preoperatively within a bowel prep regime), Norfloxacin, Levofloxacin, Sparfloxacin Antibiotics - other: Chloramphenicol, Isoniazid Antifungals: Fluconazole, Itraconazole, Ketoconazole, Posaconazole, Voriconazole Antiretrovirals: Atazanavir; Darunavir; Indinavir; Lopinavir; Nelfinavir; Ombitasvir, Paritaprevir, Ritonavir and Saquinavir. Antidepressants/ADHD: Fluvoxamine, Enoxacine. Calcium-channel blockers: Diltiazem, Verapamil Monoclonal Antibodies: Ceritinib, Idelalisib, Lonafarnib, Tucatinib. Other strong cytochrome P450 3A4 inhibitors: Cimetidine, Cobicistat; grapefruit juice, Mifepristone, Nefazodone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of disease free survival (DFS) with propofol-TIVA versus sevoflurane | Until 3 years from participant index surgery date
  The study will collect endpoint data for each participant on time of disease progression. This will be used to compare disease free survival across arms.
Comparison of disease free survival (DFS) with lidocaine compared with no lidocaine | Until 3 years from participant index surgery date
  The study will collect endpoint data for each participant on time of disease progression. This will be used to compare disease free survival across arms.

SECONDARY OUTCOMES:
Comparison of overall survival (OS) with propofol-TIVA versus sevoflurane | Until 3 years from participant index surgery date
  The study will collect endpoint data for each participant on survival status. This will be used to compare overall survival across arms.
Days alive and at home with propofol-TIVA versus sevoflurane | 30 days post surgery
  Data will be collected at thirty days post surgery regarding date of discharge from hospital and survival status. This is then used to calculate number of days alive and at home (i.e. out of hospital) and compare across arms.
Overall survival with intravenous lidocaine versus no lidocaine | Until 3 years from participant index surgery date
  The study will collect endpoint data for each participant on survival status. This will be used to compare overall survival across arms.
Days alive and at home with intravenous lidocaine versus no lidocaine | 30 days post surgery
  Data will be collected at thirty days post surgery regarding date of discharge from hospital and survival status. This is then used to calculate number of days alive and at home (i.e. out of hospital) and compare across arms.
Comparison of post-operative complications with propofol-TIVA versus sevoflurane | 5 days post surgery or at discharge if earlier
  Short term postoperative morbidity assessed by the Post Operative Morbidity Scale (POMS) with Clavien-Dindo severity grading.
  POMS is an 18-item tool that addresses nine domains of morbidity relevant to the post-surgical patient . The severity in each POMS domain will then be graded according to the Clavien-Dindo Classification on the basis of treatment applied to correct each respective complication , and captures complications within 5 grades.
Comparison of post-operative complications with intravenous lidocaine versus no lidocaine | 5 days post surgery or at discharge if earlier
  Short term postoperative morbidity assessed by the Post Operative Morbidity Scale (POMS) with Clavien-Dindo severity grading.
  POMS is an 18-item tool that addresses nine domains of morbidity relevant to the post-surgical patient . The severity in each POMS domain will then be graded according to the Clavien-Dindo Classification on the basis of treatment applied to correct each respective complication , and captures complications within 5 grades.
Comparison of chronic post surgical pain with propofol-TIVA versus sevoflurane | At 90 days and 12 months post surgery
  Pain measured using the Brief Pain Inventory Short Form. Patient reported pain on a scale of 0 to 10 where 0 is no pain and 10 is worst pain.
  Pain measured using the Neuropathic Pain Questionnaire. Patient reported neuropathic pain on a scale of 0 to 100 where 0 is no pain and 100 is worst pain.
Comparison of chronic post surgical pain with intravenous lidocaine versus no lidocaine | At 90 days and 12 months post surgery
  Pain measured using the Brief Pain Inventory Short Form. Patient reported pain on a scale of 0 to 10 where 0 is no pain and 10 is worst pain.
  Pain measured using the Neuropathic Pain Questionnaire. Patient reported neuropathic pain on a scale of 0 to 100 where 0 is no pain and 100 is worst pain.
Safety profile of propofol-TIVA versus sevoflurane | during surgery until discharge from Post Anaesthetic Care Unit (PACU) or within the first 4 hours of ICU admission
  Toxicities measured using CTCAE V 5 .0
Safety Profile intravenous lidocaine versus no lidocaine | during surgery until discharge from Post Anaesthetic Care Unit (PACU) or within the first 4 hours of ICU admission
  Toxicities measured using CTCAE V 5 .0
Concomitant medication use with propofol-TIVA versus sevoflurane | 5 days post anaesthesia
  From 2 weeks prior to surgery up to Day 5 post-surgery administration of relevant medications will be recorded
Concomitant medications use with intravenous lidocaine versus no lidocaine | 5 days post anaesthesia
  From 2 weeks prior to surgery up to Day 5 post-surgery administration of relevant medications will be recorded
Health utility with propofol-TIVA versus sevoflurane | At 30 days, 90 days and every 12 months post surgery up to 3 years
  The EQ-5D-5L is a standardised instrument for use as a measure of health outcome and is applicable to a wide range of health conditions and treatments. This five item scale covers the following dimensions (5D): mobility, self-care, usual activities, pain/discomfort and anxiety/depression, with each dimension having five levels (5L). The use of the EQ-5D-5L will enable utility valuations to be estimated for health states experienced.
Health utility with intravenous lidocaine versus no lidocaine | At 30 days, 90 days and every 12 months post surgery up to 3 years
  The EQ-5D-5L is a standardised instrument for use as a measure of health outcome and is applicable to a wide range of health conditions and treatments. This five item scale covers the following dimensions (5D): mobility, self-care, usual activities, pain/discomfort and anxiety/depression, with each dimension having five levels (5L). The use of the EQ-5D-5L will enable utility valuations to be estimated for health states experienced

OTHER OUTCOMES:
Comparison of return to intended oncological treatment (RIOT) with propofol-TIVA versus sevoflurane | At 90 days and 12 months post surgery
  Data will be collected post surgery regarding post treatment adjuvant therapy given according to plan. A comparison will be made between number of participants receiving post surgery oncological treatment as planned and the number of patients deviating from the plan in each arm of the study.
Comparison of return to intended oncological treatment (RIOT) with intravenous lidocaine versus no lidocaine | At 90 days and 12 months post surgery
  Data will be collected post surgery regarding post treatment adjuvant therapy given according to plan. A comparison will be made between number of participants receiving post surgery oncological treatment as planned and the number of patients deviating from the plan in each arm of the study.
Correlative blood studies | Preop, Day 1, 3 and 5 (if still an inpatient) and at recurrence
  Inflammatory markers - Neutrophil to lymphocyte ratio (NLR), Platelet to lymphocyte ratio (PLR), C-reactive protein (CRP) Circulating tumour deoxyribonucleic acid (ctDNA), DNA/RNA, Circulating tumour cells (CTCs), immune profile using flow cytometry and plasma for cytokines These are exploratory transnational research outcomes levels of these biomarkers will be measured over the course of the study and analysed for correlation the study outcomes.
Correlative breath biopsy studies | Preop, Day 1, 3 and 5 (if still an inpatient) and at recurrence
  To characterise the effect of anaesthetic agents on perioperative inflammatory changes will measure Targeted Volatile Organic Compounds of the eicosanoid pathway by sampling patients breath (breath biopsy) to monitor inflammatory changes within the pulmonary compartment.
MINS Substudy | Day 0 to day 30
  At sites who agree to participate:
  Blood Specimens and 12-Lead ECG - 12 Lead ECGS will be done and blood specimens collected to measure Troponin levels at baseline, Day 1 and Day 2 post op.
  Assessment of the predefined diagnostic criteria for MINS and perioperative myocardial infarction on Day 5 or Discharge if earlier Assessment of predefined diagnostic criteria for MINS and myocardial infarction at 30 days post op.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Riedel, MB.ChB, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (27):
- United States (3):
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Centre, Houston, Texas
- Australia (22):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mackay Base Hospital, Mackay, Queensland
  - RedCliffe Hospital, Redcliffe, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Ballarat Base Hospital, Ballarat Central, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Northern Hospital, Epping, Victoria
  - St Vincent's Hospital, Melbourne, Fitzroy, Victoria
  - Western Health Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Northeast Health, Wangaratta, Wangaratta, Victoria
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland

IPD SHARING:
Plan to Share IPD: No